CLINICAL TRIAL: NCT03059836
Title: Effects of n3 PUFA Supplementation on the Attenuation of Muscle Disuse Atrophy in Young Women
Brief Title: n3 PUFA and Muscle-disuse Atrophy in Young Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: University of Guelph (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1457
Record Dates: First submitted 2017-02-15; First posted 2017-02-23 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Muscle Atrophy
Keywords: n3 PUFA
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- n3 PUFA (Experimental): Intervention: n3 PUFA (3000mg of Eicosapentaenoic acid per day and 1800mg of Docosahexaenoic acid per day)
  Interventions: Dietary Supplement: n3 PUFA-enriched fish oil
- Placebo (Placebo Comparator): Intervention: Organic Sunflower Oil 5000mg per day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: n3 PUFA-enriched fish oil — 3000mg of Eicosapentaenoic acid per day and 1800mg of Docosahexaenoic acid per day
  Arms: n3 PUFA
Dietary Supplement: Placebo — Organic Sunflower Oil 5000mg per day
  Arms: Placebo

SUMMARY:
This study will examine the influence of n3 PUFA supplementation on the rate of muscle atrophy in women undergoing 2 weeks of unilateral limb immobilization. Assessments in skeletal muscle strength and skeletal muscle volume will also me made before, after and in recovery from immobilization.

DETAILED DESCRIPTION:
Biological aging is associated with the loss of skeletal muscle mass and strength resulting in compromised metabolic function and mobility. Throughout life, individuals will also experience periods of reduced physical activity/muscle disuse that independently lower muscle mass and strength accelerating the aging process. The losses in muscle mass with aging and disuse are underpinned by feeding-induced declines in rates of muscle protein synthesis. Thus, strategies to enhance muscle protein synthesis could have clinical implications for those who wish to maintain metabolic health and function during times of muscle disuse.

Supplementation with n3 PUFA-enriched fish oil has been shown to potentiate rates of muscle protein synthesis in response to simulated feeding in both younger and older adults. Fish oil supplementation also has been efficacious in enhancing skeletal muscle strength during a period of resistance exercise training. However, no study has examined the impact of fish oil supplementation to enhance muscle protein synthesis and offset declines in muscle mass/strength during a period of immobilization.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 18-30 years

Exclusion Criteria:

* Take any analgesic or anti-inflammatory drugs(s), prescription or non-prescription, chronically will be excluded
* A history of neuromuscular problems or muscle and/or bone wasting diseases
* Any acute or chronic illness, cardiac, pulmonary, liver, or kidney abnormalities, uncontrolled hypertension, insulin- or non-insulin dependent diabetes or other metabolic disorders-all ascertained through medical history screening questionnaires
* Use medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories, or prescription strength acne medications)
* Fish allergy

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self-representation of gender identity
Enrollment: 20 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Muscle Volume | Baseline (0 days), After (14 days) of unilateral limb immobilization and at 14 days post immobilization
  Change in Muscle Volume Measured by Magnetic Resonance Imaging

SECONDARY OUTCOMES:
Integrated Rates of Muscle Protein Synthesis | Before (0 days), During (0-14 days inclusive), and After (14-28 days inclusive) of unilateral limb immobilization
  Change in Muscle Protein Synthesis
Skeletal Muscle Strength | Before (0 days), After (14 days) of unilateral limb immobilization and at 14 days Post immobilization
  Change in Skeletal Muscle Strength
Muscle Lipid Composition | Baseline (-28 days), and at Before (0 days), After (14 days) of unilateral limb immobilization and at 14 days Post immobilization
  Change in Muscle Lipid Composition

CONTACTS AND LOCATIONS:
Overall Officials: Stuart M Phillips, PhD, Principal Investigator — McMaster University
Locations (1):
- Exercise Metabolism Research Laboratory, McMaster Univeristy, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No